CLINICAL TRIAL: NCT05606146
Title: Phase IIc (Protocol 55P127): Addition of up to 10 Women to Explore Silver Systemic Absorption as a Continuation Study to: Phase IIb (Protocol 55P140)
Brief Title: IUB SEAD RED (Revolutionary Endometrial Ablation Device Study)
Acronym: HMB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ocon Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 55P127
Record Dates: First submitted 2022-10-24; First posted 2022-11-04 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Heavy Menstrual Bleeding
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Intervention Model Description: Endometrium ablation with the IUB SEAD device
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): IUB SEAD procedure
  Interventions: Device: IUB SEAD

INTERVENTIONS:
Device: IUB SEAD — The investigative device, the IUB SEAD™, is a novel spherical endometrial ablation device developed to allow for simple, office-based chemical EA to treat benign causes of the symptom of HMB

SUMMARY:
One of the AUB symptoms, heavy menstrual bleeding (HMB), can lead to iron deficiency and iron deficiency anemia and in acute and severe cases, can necessitate emergency medical care. This study's focus is on the symptom of HMB which has a number of benign causes.

The investigative device, the IUB SEAD™, is a novel spherical endometrial ablation device developed to allow for simple, office-based chemical EA to treat benign causes of the symptom of HMB. The suggested procedure is expected to be simpler than the currently available EA methods and yet should still reduce the need for a hysterectomy.

DETAILED DESCRIPTION:
Chronic abnormal uterine bleeding (AUB), involving menstrual bleeding of abnormal quantity, duration, frequency, or regularity is experienced by 10-50% of women of reproductive age, adversely impacts quality of life, and can have substantial adverse economic impacts on patients, and healthcare systems. One of the AUB symptoms, heavy menstrual bleeding (HMB), can lead to iron deficiency and iron deficiency anemia and in acute and severe cases, can necessitate emergency medical care. This study's focus is on the symptom of HMB which has a number of benign causes.

While pharmacologic treatment options exist, they are not always effective, and they are frequently associated with both side effects and ongoing cost of care. Consequently, some women desire more definitive options. Endometrial ablation (EA) is a minimally invasive approach designed to manage a number of the causes of HMB and can be performed under direct intrauterine vision with resectoscopic instruments or with a non-resectoscopic approach (non-resectoscopic endometrial ablation or NREA). For NREA, one of a number of specially designed device is inserted into the endometrial cavity to deliver thermal, cryogenic or radiofrequency electrical energy in an attempt to destroy the uterine lining or endometrium. In some jurisdictions, NREA has become an accepted office-based procedure, but is still usually performed in an institutional setting, is associated with risks associated with the procedure, anesthesia, and subsequent infertility, and has a failure rate that averages about 26%. These devices are typically expensive and require training for the surgeon and the ancillary support staff.

The investigative device, the IUB SEAD™, is a novel spherical endometrial ablation device developed to allow for simple, office-based chemical EA to treat benign causes of the symptom of HMB. The suggested procedure is expected to be simpler than the currently available EA methods and yet should still reduce the need for a hysterectomy. This study will evaluate an additional exploratory endpoint in order to evaluate if there are detectable levels of silver in blood following SEAD treatment. SEAD treatment is performed locally by intrauterine administration for a duration of 30 minutes, during which the silver nitrate beads gradually dissolve. Upon dissolution the silver ions act on the mucus layer of the endometrium by binding to proteins and causing their denaturation, resulting in the formation of an eschar. The effect is local, and the bound silver is no longer active therefore it is unlikely that 100% of the silver dose will be available for absorption.

ELIGIBILITY:
Inclusion Criteria:

1. Female subject age 40 to 50 years, inclusive
2. Suffering from the symptom of heavy menstrual bleeding (HMB) from benign causes with no definable organic cause and are candidates for endometrial ablation or surgical treatment.
3. PBAC score of >150 - an average of 2 consecutive screening scores prior to study treatment
4. Are thought to be ovulatory with cyclic predictable onset of menses with a cycle length of 24-38 days.
5. Have either a normal appearing endometrial cavity as assessed by hysteroscopy performed within 90 days of study treatment, or one that is distorted by a FIGO Type 2 submucous leiomyoma ≤3 cm in mean diameter.
6. Have endometrial sampling with normal histology within 6 months of the study procedure.
7. Premenopausal status confirmed by FSH level measurement at screening (FSH < 40 IU/L). FSH level measurement will be repeated in case of a borderline result
8. Screening hemoglobin levels >9.0 g/dL
9. Uterine sound measurement of 6.5-12 cm (external os to internal fundus)
10. Negative serum pregnancy test at the Screening visit and on the day of SEAD™ treatment
11. women whose sexual activity places them at risk for pregnancy must agree to use an effective, non-hormonal, non-intrauterine method of contraception throughout the course of the study. For this study, acceptable effective methods of contraception are considered to be those listed below:

    * Barrier method, i.e., (a) condom (male or female) with spermicide or (b) diaphragm with spermicide or
    * Vasectomy (partner), or
    * Abstinence, if in line with the preferred and usual lifestyle of the subject [where abstinence is defined as refraining from heterosexual intercourse]
12. Subject is able to understand and sign a written informed consent form
13. Subject is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
14. The subject demonstrates an understanding of how to record menstrual blood loss using a menstrual pictogram

Exclusion Criteria:

1. Pregnant women or those who desire to conceive at any time in the future
2. An endometrial cavity with any of the following: congenital malformation of (eg septate uterus), endometrial polyp >8 mm in largest dimension, FIGO Type 0 or 1 leiomyomas of any diameter or Type 2 leiomyomas > 3 cm in mean diameter; intrauterine adhesions/ synechiae that distort the endometrial cavity sufficient to impair deployment of the SEAD device.
3. Underwent prior uterine surgery that interrupts the integrity of the uterine wall (e.g., transmural abdominal (laparoscopic or laparotomic) or hysteroscopic myomectomy and/or metroplasty during last 3 months prior to screening, classical Cesarean section, or endometrial ablation
4. Have an abnormal endometrial biopsy that suggests either anovulation or a risk for the development of endometrial cancer (i.e., benign hyperplasia, endometrial hyperplasia with atypia, endometrial intraepithelial neoplasia, endometrial cancer)
5. Have a documented clinical history of titanium allergy or hypersensitivity to any component of IUB™SEAD™.
6. Suffers from active endometritis, active pelvic inflammatory disease (PID) or active sexually transmitted disease (STD)
7. Suffers from active infection of the genitals, vagina, cervix, or uterus
8. Presence of bacteremia, sepsis, or other active systemic infection
9. Known/suspected abdominal, pelvic, or gynecological malignancy within the past 5 years
10. Known clotting defects or bleeding disorders
11. Currently using anticoagulant treatment
12. Subjects with abnormal Papanicolaou (Pap) test or atypical squamous cells of undetermined significance (ASCUS) with positive high-risk human papilloma virus (HPV) test result within the appropriate screen timeframe, and prior to SEAD™ treatment. Alternatively, a colposcopy performed prior to SEAD™ treatment, that showed evidence of dysplasia requiring treatment. In case treatment was performed > 6 months prior to enrollment and follow-up was done with no evidence of disease by clinical evaluation, the subject is eligible.
13. Suffers from clinically significant adenomyosis indicated by subject complaints or imaging
14. Presence of an implantable contraceptive device, unless subject agrees to have the device removed immediately on screening, and prior to PBLAC assessment
15. Post-partum ≤ 6-months
16. Currently participating in or considering participation in a research study of an investigational drug or device that would begin during the course of this investigational study
17. Any general health or mental, or other situation or condition which, in the opinion of the Investigator, could present an increased risk for the subject or impact the subject's ability to comply with protocol requirements.
18. Has a polyp that was not removed before day of treatment

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Gender having a uterus
Enrollment: 10 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence and characteristics of device and/or procedure related adverse events (AEs) | 6 months
  occurring during the 6-months following SEAD™ device treatment
Efficacy: Change in bleeding volume | 6 months
  measured by Pictorial Blood Loss Assessment Chart (PBAC) at 6 months post-treatment compared to baseline.

SECONDARY OUTCOMES:
Change from baseline quality of life (QoL) | 36 months
  as assessed using the MIQ questionnaire at 6, 12, 24- and 36-months post-treatment.
Change in bleeding volume | 36 months
  measured by Pictorial Blood Loss Assessment Chart (PBAC) at 12, 24- and 36-months post treatment.

OTHER OUTCOMES:
SEAD levels in blood at baseline | 3 months
  (prior to treatment) and at 1, 2 hours following treatment (post insertion), and at 1 day, 7 days, and 3 months following treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Noam Smorjick, MD, Principal Investigator — Shamir medical center ,Rishon LeZion
Locations (1):
- Shamir medical center, Rishon LeZiyyon, Israel

IPD SHARING:
Plan to Share IPD: No